CLINICAL TRIAL: NCT05317507
Title: Safety of Co-Administered CHI-554 and Alcohol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Sara K Blaine, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 710022US1313
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: During the Experimental portion of the study, participants will be randomized to a dosing order of 3 different doses. During the at-home portion of the study all participants will receive the same dose for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experimental portion of the study is double blind.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Randomization order 1 (Experimental): Participants receive placebo at visit 1, 50 mg CBD at visit 2, and 100 mg CBD at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo
- Randomization order 2 (Experimental): Participants receive placebo at visit 1, 100 mg CBD at visit 2, and 50 mg CBD at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo
- Randomization order 3 (Experimental): Participants receive 50 mg CBD at visit 1, placebo at visit 2, and 100 mg CBD at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo
- Randomization order 4 (Experimental): Participants receive 50 mg CBD at visit 1, 100 mg CBD at visit 2, and placebo at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo
- Randomization order 5 (Experimental): Participants receive 100 mg CBD at visit 1, 50 mg CBD at visit 2, and placebo at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo
- Randomization order 6 (Experimental): Participants receive 100 mg CBD at visit 1, placebo at visit 2, and 50 mg CBD at visit 3 followed by a 4-week period of at home use of 100 mg CBD daily.
  Interventions: Drug: CBD oil; Drug: Placebo

INTERVENTIONS:
Drug: CBD oil — 50 mg
Drug: CBD oil — 100 mg CBD
Drug: Placebo — Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind study to assess the safety, tolerability, and effects of CHI-554 when co-administered with alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy adult aged 21-65 years, inclusive, at the time of screening.
* Has a body mass index between 18 and 35 kg/m2 (inclusive).
* Reports at online screening (and confirmed at in-person screening) that has achieved a calculated blood alcohol concentration of at least .06% in the past month according to the Daily Drinking Questionnaire (Collins et al., 1985).
* Is judged by the Investigator to be in generally good health at screening based on participants' medical history, vital signs, and comprehensive metabolic panel test results. Laboratory results outside of the reference range but within acceptable limits must be documented as not clinically significant (NCS) at the discretion of the Investigator.
* Must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.
* Able to read and write in English.

Exclusion Criteria:

* Women who are pregnant, lactating, breastfeeding, or planning a pregnancy.
* Women of childbearing potential who are unwilling or unable to use an acceptable method of contraception (abstinence or the use of a highly effective method of contraception, including hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, vasectomy, or intrauterine device) from at least 21 days prior to the first dose of study medication until 28 days after the last dose of study medication.
* Has a history of epilepsy, hepatitis, clinically significant hepatic or renal impairment, or human immunodeficiency virus.
* Changes in the use of a prescription, over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) for 28 days prior to the Screening Visit.
* Current use of any known hepatotoxic medication.
* Has any clinically significant condition or abnormal finding at screening that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study IP.
* Has a history of a known significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to cannabis, including phytocannabinoids and cannabinoid analogues, or excipients utilized within the IP (e.g., coconut; coconut oil; medium-chain triglycerides).
* Has taken a medication with likely CBD-interactions, including warfarin, clobazam, valproic acid, phenobarbital, mTOR inhibitors, oral tacrolimus, and St. John's Wort within 28 days of the Screening Visit or during the study.
* Has taken grapefruit products and/or Seville oranges within the 7 days prior to the first Experimental Visit.
* Has used cannabis, synthetic cannabinoid or cannabinoid analogues (e.g., dronabinol, nabilone), hemp products, synthetic cannabinoid receptor agonists (e.g., Spice, K2), or any CBD- or THC-containing product (e.g., Sativex, Epidiolex) within 28 days of the Screening Visit or during the study.
* Has a past or current severe Alcohol Use Disorder as assessed by the Structured Clinical Interview Diagnostic (SCID) for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) at the Screening Visit.
* Has a past or current diagnosis of a significant psychiatric disorder, or current use of illicit drugs, as assessed by the SCID at the Screening Visit that would, in the opinion of the Investigator, affect the subject's ability to comply with the study requirements.
* Endorses current suicidal intent as assessed by the SCID at the Screening Visit.
* Has participated in any investigational product or device study within 30 days prior to the Screening Visit, or is scheduled to participate in another investigational product or device study during the course of this study.
* Demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.
* Has a positive result on an alcohol breath test or urine drug screen for benzodiazepines, PCP, barbiturates, antidepressants, cocaine, amphetamine, methamphetamine, THC, and opiates at the Screening Visit or at any Experimental Visit.
* Self-reports current use of nicotine-containing products or nicotine replacement products as assessed by the SCID at the Screening Visit.
* Anyone with a history of hypersensitivity to cannabidiol will not be enrolled in the study. - To avoid any potential drug-drug interactions, participants must not be taking any of the following at any time during study participation: CYP3A4 or CYP2C19 Inducers, CYP1A2, CYP2B6, CYP2C8, CYP2C9, and CYP2C19 Substrates (e.g.,, theophylline, or tizanidine), CYP2B6 substrates (e.g., bupropion, efavirenz), uridine 5'-diphospho-glucuronosyltransferase 1A9 (UGT1A9) substrates (e.g., diflunisal, propofol, fenofibrate), and UGT2B7 substrates (e.g., gemfibrozil, lamotrigine, morphine, lorazepam), CYP2C8 and CYP2C9 (e.g., phenytoin) substrates, drugs that are metabolized by (i.e., are substrates of) CYP2C19 (e.g., diazepam), stiripentol, everolimus, sirolimus, tacrolimus, digoxin, and Valproate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events/Serious Adverse Events | Day 0
  Adverse Events/Serious Adverse Events
Adverse Events/Serious Adverse Events | Day 3
  Adverse Events/Serious Adverse Events
Adverse Events/Serious Adverse Events | Day 6
  Adverse Events/Serious Adverse Events
Adverse Events/Serious Adverse Events | Day 34
  Adverse Events/Serious Adverse Events
Change from baseline in Alanine aminotransferase (ALT) | Day 0
  Alanine aminotransferase (ALT)
Change from baseline in Alanine aminotransferase (ALT) | Day 3
  Alanine aminotransferase (ALT)
Change from baseline in Alanine aminotransferase (ALT) | Day 6
  Alanine aminotransferase (ALT)
Change from baseline in Alanine aminotransferase (ALT) | Day 34
  Alanine aminotransferase (ALT)
Change from baseline in blood pressure | Day 0
  Blood pressure (systolic and diastolic)
Change from baseline in blood pressure | Day 3
  Blood pressure (systolic and diastolic)
Change from baseline in blood pressure | Day 6
  Blood pressure (systolic and diastolic)
Change from baseline in blood pressure | Day 34
  Blood pressure (systolic and diastolic)

SECONDARY OUTCOMES:
Peak Blood Alcohol Level (BAL) | Day 0
  Peak BAL during experimental visits
Peak Blood Alcohol Level (BAL) | Day 3
  Peak BAL during experimental visits
Peak Blood Alcohol Level (BAL) | Day 6
  Peak BAL during experimental visits

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States